CLINICAL TRIAL: NCT04202653
Title: New Combination of ETV, TQ-A3334 and TQ-B2450 for the Treatment of Chronic Hepatitis B Virus Infection
Brief Title: Combination of ETV, TQ-A3334 and TQ-B2450 for CHB (Neptune Study)
Acronym: Neptune
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qin Ning, Director, Head of Department of Infectious Diseases, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQ-A3334-II-02
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Naive:ETV (Active Comparator): Entecavir 0.5 mg po daily for 24 weeks in naive patients
  Interventions: Drug: ETV
- Naive:ETV+TQ-A3334 (Experimental): Entecavir 0.5 mg po daily plus TQ-A3334 for 24 weeks in naive patients
  Interventions: Drug: ETV; Drug: TQ-A3334
- Naive:ETV+TQ-A3334+TQ-B2450 (Experimental): Entecavir 0.5 mg po daily plus TQ-A3334 plus inhibitor of TQ-B2450 for 24 weeks in naive patients
  Interventions: Drug: ETV; Drug: TQ-A3334; Drug: TQ-B2450
- Experienced:ETV (Active Comparator): Entecavir 0.5 mg po daily for 24 weeks in treatment experienced patients
  Interventions: Drug: ETV
- Experienced:ETV+TQ-A3334 (Experimental): Entecavir 0.5 mg po daily plus TQ-A3334 for 24 weeks in treatment experienced patients
  Interventions: Drug: ETV; Drug: TQ-A3334
- Experienced:ETV+TQ-A3334+TQ-B2450 (Experimental): Entecavir 0.5 mg po daily plus TQ-A3334 plus TQ-B2450 for 24 weeks in treatment experienced patients
  Interventions: Drug: ETV; Drug: TQ-A3334; Drug: TQ-B2450

INTERVENTIONS:
Drug: ETV — entecavir 0.5 mg qd
Drug: TQ-A3334 — TQ-A3334 po qw
  Arms: Experienced:ETV+TQ-A3334; Experienced:ETV+TQ-A3334+TQ-B2450; Naive:ETV+TQ-A3334; Naive:ETV+TQ-A3334+TQ-B2450
Drug: TQ-B2450 — TQ-B2450 q3w iv
  Arms: Experienced:ETV+TQ-A3334+TQ-B2450; Naive:ETV+TQ-A3334+TQ-B2450

SUMMARY:
This study is a single-center, randomized, prospective, open-label Phase 2 Clinical trial to evaluate efficacy and safety of ETV and TQ-A3334 combinated with/without inhibitor of TQ-B2450 versus ETV alone in chronic hepatitis B patients. Patients were randomized to one of 3 different antiviral treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients from 18 to 65 years of age;
2. Chronic hepatitis B infection
3. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug;
4. Agree to participate in the study and sign the patient informed consent.

Exclusion Criteria:

1. Patients who had NAs resistance;
2. Other antiviral, anti-neoplastic or immunomodulatory treatment;
3. Women with ongoing pregnancy or breast-feeding;
4. Co-infection with active hepatitis A, hepatitis C, hepatitis D(Those hospitals which have the ability to do the test will do) and/or human immunodeficiency virus (HIV);
5. ALT >10 ULN;
6. LSM >9kPa ;
7. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia);
8. Signs or symptoms of hepatocellular carcinoma;
9. Neutrophil count < 1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening;
10. Hemoglobin < 11.5 g/dL for females and <12.5 g/dL for men;
11. Serum creatinine level > 1.5 ULN in screening period.
12. Phosphorus < 0.65 mmol/L;
13. ANA > 1:100;
14. History of severe psychiatric disease;
15. History of a severe seizure disorder or current anticonvulsant use;
16. History of immunologically mediated disease, (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.);
17. History of chronic pulmonary disease associated with functional limitation;
18. Diseases that IFN and Nucleotides or nucleosides are not suitable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HBsAg quantification at week 24 | week 24
  HBsAg quantification are measured

SECONDARY OUTCOMES:
HBsAg loss rates at week 24 | week 24
  HBsAg loss rates are measured
HBsAg seroconversion rates at week 24 | week 24
  HBsAg seroconversion rates are measured
HBeAg loss rates at week 24 | week 24
  HBeAg loss rates are measured
HBeAg seroconversion rates at week 24 | week 24
  HBeAg seroconversion rates are measured
HBV DNA<20IU/mL rates at week 24 | week 24
  HBV DNA<20IU/mL rates are measured